CLINICAL TRIAL: NCT07310524
Title: A Randomized Double-Blind Controlled Trial Comparing Opioid-Free Anesthesia and Opioid-Based Anesthesia on the qNOX Index During Abdominal Surgery Under General Anesthesia
Brief Title: COMPARISON OF OPIOID-FREE AND OPIOID-BASED ANESTHESIA TECHNIQUES ON qNOX INDEX IN ABDOMINAL SURGERY UNDER GENERAL ANESTHESIA
Acronym: OFA-OBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Rahman Efendi Nasution (Other)
Responsible Party: Sponsor-Investigator, Muhammad Rahman Efendi Nasution, Sponsor-Investigator (Principal Investigator), Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRENST2025
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Opioid-free Anesthesia
Keywords: opioid-free anesthesia, opioid-based anesthesia, qNOX, abdominal surgery
MeSH Terms: interventions — Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: This study uses a randomized parallel assignment design in which participants are allocated into two groups: an opioid-free anesthesia (OFA) protocol group and an opioid-based anesthesia (OBA) protocol group. Each participant receives only one assigned anesthetic protocol throughout the surgical procedure. The model allows comparison of postoperative pain scores, opioid consumption, and recovery outcomes between the two independent groups.
Masking Description: Participants and all clinical staff involved in intraoperative management, including anesthesia providers and outcome assessors, were blinded to group allocation. Drug preparation and labeling were performed by an independent pharmacist who was not involved in patient care or data collection. Study medications were placed in identical syringes to maintain blinding throughout the perioperative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine for sedation and sympatholysis, low-dose ketamine for analgesia and prevention of ce (Experimental): Participants in this arm will receive opioid-free anesthesia (OFA), an anesthetic technique that avoids the use of intraoperative opioids and employs a multimodal non-opioid regimen. The protocol includes agents such as dexmedetomidine, low-dose ketamine, intravenous lidocaine, magnesium sulfate, acetaminophen, and nonsteroidal anti-inflammatory drugs (NSAIDs), administered according to institutional protocols to provide adequate anesthesia and analgesia while minimizing opioid exposure.
  Interventions: Drug: Non Opioid Analgesics
- fentanyl or remifentanil, administered according to institutional protocols (Experimental): Participants in this arm will receive opioid-based anesthesia (OBA), the standard anesthetic technique using intraoperative opioids such as fentanyl or remifentanil, administered according to institutional protocols. This arm serves as the active comparator for evaluating differences in postoperative outcomes compared with opioid-free anesthesia.
  Interventions: Drug: Non Opioid Analgesics

INTERVENTIONS:
Drug: Non Opioid Analgesics — Participants in this arm will receive opioid-free anesthesia (OFA), an anesthetic approach that avoids the use of intraoperative opioids and utilizes a multimodal non-opioid regimen. The protocol includes dexmedetomidine for sedation and sympatholysis, low-dose ketamine for analgesia and prevention of central sensitization, intravenous lidocaine for systemic analgesic and anti-inflammatory effects, magnesium sulfate as an N-methyl-D-aspartate (NMDA) receptor antagonist to enhance analgesia, acetaminophen for central non-opioid analgesia, and nonsteroidal anti-inflammatory drugs (NSAIDs) for peripheral analgesic and anti-inflammatory effects. These agents are administered according to institutional protocols to provide adequate anesthesia and analgesia while minimizing opioid exposure.

SUMMARY:
This study is a randomized, double-blind controlled clinical trial designed to evaluate the effects of opioid-free anesthesia (OFA) compared with opioid-based anesthesia (OBA) in adult patients undergoing elective abdominal surgery under general anesthesia. Opioid-free anesthesia uses a multimodal combination of ketamine, lidocaine, and dexmedetomidine to provide analgesia and autonomic stability without intraoperative opioid administration. In contrast, the opioid-based approach utilizes fentanyl as the primary analgesic agent, which remains the conventional method in many surgical settings.

The primary objective of this study was to compare the nociceptive response between OFA and OBA techniques using the qNOX index, a quantitative parameter provided by the CONOX® monitor that reflects the probability of patient response to noxious stimuli. qNOX values were recorded at several key intraoperative time points: before induction, during intubation, before incision, during the surgical incision, and one hour after incision. Secondary outcomes included intraoperative hemodynamic stability and the incidence of postoperative nausea and vomiting (PONV).

A total of 42 patients were enrolled and randomly assigned into two equal groups. Both groups underwent surgery under standardized protocols to ensure comparable anesthetic depth and surgical conditions. The study found no significant differences in qNOX values between the OFA and OBA groups at any measured time point, suggesting that nociceptive control was equally effective in both techniques. Hemodynamic parameters remained stable and comparable across groups throughout the intraoperative period.

However, a notable difference was observed in the incidence of postoperative nausea and vomiting. The OFA group experienced a significantly lower rate of PONV compared to the OBA group, indicating a potential clinical benefit of avoiding intraoperative opioid exposure. These findings support the use of OFA as a safe and effective alternative to traditional opioid-based strategies, particularly in patients at risk for opioid-related adverse effects.

Overall, this study provides evidence that opioid-free anesthesia can offer equivalent intraoperative analgesic control while reducing postoperative opioid-associated complications.

DETAILED DESCRIPTION:
Opioid-based anesthesia has long been the standard approach for providing analgesia and autonomic stability during general anesthesia. However, increasing awareness of opioid-related adverse effects such as respiratory depression, postoperative nausea and vomiting (PONV), delayed recovery, hyperalgesia, and risks of prolonged opioid exposure has led to the development of alternative strategies that aim to reduce or eliminate the use of intraoperative opioids. Opioid-free anesthesia (OFA) is one such technique that utilizes a multimodal combination of non-opioid agents to achieve adequate analgesia and hemodynamic control while minimizing the pharmacologic burden associated with opioids.

OFA protocols typically incorporate medications such as ketamine, lidocaine, and dexmedetomidine, each contributing analgesic, antihyperalgesic, and sympatholytic effects through different mechanisms. This multimodal approach may offer more stable nociceptive control and reduce the incidence of opioid-related postoperative complications. Despite these potential benefits, evidence comparing OFA and traditional opioid-based anesthesia (OBA) in terms of intraoperative nociceptive response remains limited, particularly when assessed using objective monitoring systems.

The present study was designed as a randomized, double-blind controlled clinical trial to evaluate whether OFA provides comparable intraoperative nociceptive control to OBA in patients undergoing elective abdominal surgery under general anesthesia. The nociceptive response was assessed using the qNOX index, a quantitative parameter derived from electroencephalographic and electromyographic signals provided by the CONOX® monitoring system. qNOX reflects the probability of patient responsiveness to noxious stimuli, offering an objective measure of intraoperative analgesic adequacy.

A total of 42 adult patients meeting the inclusion criteria were randomly assigned into two equal groups: the OFA group and the OBA group. Both groups underwent a standardized anesthetic induction and maintenance protocol to ensure comparable levels of hypnosis and neuromuscular blockade. The OFA group received a combination of ketamine, lidocaine, and dexmedetomidine, while the OBA group received fentanyl as the primary opioid analgesic. All other anesthetic components, including induction agents, maintenance agents, ventilation parameters, and surgical procedures, were kept consistent between groups.

qNOX values were recorded at predetermined intervals representing key phases of the surgical process: baseline prior to induction, during endotracheal intubation, prior to surgical incision, at the moment of incision, and one hour following incision. Hemodynamic parameters were monitored throughout the procedure to evaluate autonomic stability. In addition to nociceptive monitoring, postoperative outcomes including nausea, vomiting, and overall recovery quality were assessed in the postoperative care unit.

This study seeks to determine whether OFA can provide an intraoperative nociceptive profile comparable to OBA, while potentially reducing postoperative opioid-related adverse effects. The findings are expected to contribute to the growing body of evidence regarding the clinical utility, safety, and feasibility of implementing opioid-free anesthesia in routine surgical practice, particularly for patients at higher risk of opioid-related complications.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged 18-65 years

Patients undergoing elective abdominal surgery (e.g., laparotomy, colectomy, cystectomy, etc.)

American Society of Anesthesiologists (ASA) physical status I-II

Undergoing general anesthesia with endotracheal intubation

Undergoing abdominal surgery with a duration of less than 4 hours

Willing to participate in the study and sign the informed consent form

Patients who are extubated in the operating room after completion of the surgical procedure

Exclusion Criteria:

Patients with neurological disorders (e.g., epilepsy, stroke, altered level of consciousness)

History of severe psychiatric disorders or long-term use of psychotropic medications

Patients with a history of cardiac arrhythmias and/or prior use of antiarrhythmic drugs and/or those with a pacemaker

Patients with increased intracranial pressure

Patients on chronic opioid therapy or other chronic pain treatments

Patients with severe hemodynamic instability (hypotension/shock, unstable arrhythmias)

Patients with a history of allergy to medications used in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Time to Extubation | Immediately postoperative (0-30 minutes)
  Time (in minutes) measured from the discontinuation of general anesthetic agents until successful extubation in the operating room. The measurement reflects the patient's recovery speed from anesthesia following elective abdominal surgery performed under general anesthesia with endotracheal intubation.

SECONDARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-24 hours postoperatively
  The proportion of patients who experience postoperative nausea and/or vomiting within the early postoperative period following abdominal surgery under general anesthesia. Assessment will be performed using direct clinical observation and patient self-reporting in the recovery area.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUP H. Adam Malik Medan, Medan, North Sumatra, Indonesia